CLINICAL TRIAL: NCT03041571
Title: Patients to People: Examining the Effects of Early Implementation of Narrative Medicine Techniques on Patient Centered Attitudes in Medical Students. A Qualitative Study
Brief Title: Impact of Early Implementation of Narrative Medicine Techniques on Patient Centered Attitudes of Medical Students
Status: Withdrawn | Type: Observational
Why Stopped: PI is no longer with UF. No New PI assigned to date.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201601597
Record Dates: First submitted 2017-01-31; First posted 2017-02-02 (Estimated); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Narrative Medicine; Chronic Disease; Terminal Illness; Cancer; Diabetes Mellitus; Cystic Fibrosis; Rheumatologic Disorder; Oncologic Disorders; Hematologic Diseases
MeSH Terms: conditions — Narrative Medicine; Chronic Disease; Neoplasms; Diabetes Mellitus; Cystic Fibrosis; Collagen Diseases; Hematologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medical Honors Students: The Medical Honors Program students will fill out the Patient Provider Orientation Scale (PPOS). MHP students will then interview a patient with a chronic or life limiting illness.
  Interventions: Behavioral: Patient Provider Orientation Scale; Behavioral: Interview performed by MHP student
- Patients with chronic illnesses: The patients will fill out the PPOS scale. The patient will then have an Interview performed by MHP student
  Interventions: Behavioral: Patient Provider Orientation Scale; Behavioral: Interview performed by MHP student

INTERVENTIONS:
Behavioral: Patient Provider Orientation Scale — Investigators are interested in the impact that our activity has on the students' patient-centeredness. Investigators will use the Patient-Practitioner Orientation Scale (PPOS), which will be completed by both the student and the patient prior to the encounter. Following the interview, the co-investigators will lead a discussion with the patient and student. Investigators will discuss differences in patient and student PPOS scores, and how each party felt the interview went. Investigators will examine if the patients feel the interview differed from typical interactions with health care providers, and how this made the patient feel. The students will describe what was learned from the patients story as well as try to explore reasons why providers may not always learn the patient's illness story.
Behavioral: Interview performed by MHP student — The MHP students took a course called Medical Humanities in the fall of 2016. MHP students learned patient interviewing skills and the importance of gathering the patients "illness story". The students will conduct an interview with a patient with chronic illness, which will be focused on gather information about how the patients illness affects daily life as well as interactions with the health care system.

SUMMARY:
A qualitative study assessing the impact of early narrative medicine practice on Medical Honors Program (MHP) students' attitudes regarding patient-centered interactions, through interviewing patients with chronic or life-limiting illnesses to obtain their illness stories.

MHP students will develop a patient narrative for the patients interviewed. These narratives will be edited by the patient, and, with the permission of the patients, may be published as a collection of stories.

DETAILED DESCRIPTION:
Teach MHP Students about obtaining the illness story and narrative medicine. This will be done during the curriculum of the Medical Humanities class in the fall of 2016.

Recruit patients on units and floors in Shands University of Florida (UF) Health that may potentially have patients that will be good candidates for enrollment in the patient narratives. These may include pediatric hematology and oncology patients, adult hematology and oncology patients, patients with diabetes, organ transplant patients, cystic fibrosis patients, and rheumatologic disorder patients. Investigators will communicate with child life/social workers, as well as faculty medical providers on these inpatient services to help identify appropriate patients for referral and recruitment. These faculty members will obtain authorization from the patient for the investigators to approach the patient regarding recruitment.

Once a patient has been identified, a co-investigator will introduce the project to the patient, review examples of the types of questions to be asked by the MHP student, provide opportunity for questions, obtain informed consent, and provide them with the patient-practitioner orientation scale (PPOS) for completion.

A MHP student will meet with the co-investigator, fill out the PPOS, and then interview the patient. The co-investigator will be present for the interview, but the investigator would like the MHP student to conduct the interview. The interview will be voice recorded with encryption for later transcription.

Following the interview, a co-investigator will lead a discussion to determine patient and student observations/opinions about such conversations. The co-investigator will address differences in PPOS responses from patient vs student, without specifically revealing the personal answers of each, and allow for discussion of how scales can be aligned to better the patient-physician relationship. This discussion will be voice recorded for transcription and qualitative analysis by the investigators

Following the interview, the MHP students will transcribe the patient narrative. During the interview, the student and patient will agree on whether the narrative is written from the first or third person point of view.

The initial informed consent will have a specific series of check boxes to address whether the patient approves of dissemination of their story. This initial consent will specifically state that this narrative will not be published prior to their approval of the final product. The patient will also have the opportunity to declare which patient identifiers, if any, will be changed for the publication. The narrative will be presented to the patient, who will then have the opportunity to make changes and edits. If extensive edits are necessary, a subsequent narrative will be presented to the patient for final approval prior to publication. The investigators will make every effort to get the patient approval in person, however because of the possibility of the patient being discharged before the narrative has been composed, investigators will identify an acceptable method of communication with the patient outside of the hospital (email, phone call) for this purpose. In the case of the patient being discharged and needing to obtain approval, verbal approval over the phone will be obtained by a co-investigator and a witness, and will keep this documentation in a binder locked in the PI's office.

Following the completion of the interviews, the MHP students will meet for a focus group to discuss as a group their observations from their patient encounters. This focus group will be audio recorded and transcribed by the co-investigators for qualitative analysis

After all patient narratives have been completed, narratives may be published in an online or book format, following the consent that the patient provided.

ELIGIBILITY:
Inclusion Criteria:

* Patient inclusion criteria:

  * Patient of Shands UF Health or Shands Children's hospital
  * Children must be at least 8 years old
  * Patients diagnosed with chronic or potentially life-limiting illnesses
  * Patients must be English speaking
* Student Inclusion criteria

  * UF students enrolled in the Medical Honors Program
  * Medical Honors students must be up to date on HIPAA training and Confidentiality statement agreement
  * Students must take the Medical Humanities course
  * UF college of medicine students

Exclusion Criteria:

* Patient exclusion criteria:

  * Anyone that the medical social worker or Child life specialist feels would be unwilling or unable to participate in the study
  * Patients who at the time of interview are unfit to communicate (ex. Ventilated, comatose)
  * Patients less than eight years old
  * Patients that do not speak English
* Student exclusion criteria:

  * Students not enrolled in the UF College of Medicine
  * Students not enrolled in the Medical Humanities course

Ages: 8 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study population is two-fold. First the MHP students will be recruited and consented. Their participation is voluntary and will not affect their grades. Second, patients will be recruited based on the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-18 (Actual)

PRIMARY OUTCOMES:
Patient provider orientation scale score (PPOS) | baseline
  The PPOS is an 18 item questionnaire developed to evaluate patient centered care. The items are rated on a 6 point Likert-type scale. It has two separate parts, sharing and caring, that can be either summed or divided for scoring purposes. Higher scores indicate more patient centeredness.

SECONDARY OUTCOMES:
Patient provider orientation scale- "Sharing" portion | baseline
  Total from the questions related to "sharing" on the PPOS. The sharing portion relates to how open the provider is in sharing power in the patient-physician relationship, or in the case of the patient filling out the form, how much the patient wishes to share the power in the patient-physician relationship.
Patient provider orientation scale- "Caring" portion | baseline
  Total from the questions related to "caring" on the PPOS. The caring portion relates to how oriented the provider is in caring for the patient as a person and not just a disease.
Patient and Student post-interview discussion | immediately post-interview, up to 1 day
  qualitative measurement of topics and themes discussed in immediate post-interview discussion between the co-investigator, MHP student, and patient
Medical honors students focus group | following completion of all MHP/Patient interviews, up to 4 months
  qualitative measurement of topics and themes discussed in the focus group held following all MHP students completing their individual interviews

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lawrence, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Batt-Rawden SA, Chisolm MS, Anton B, Flickinger TE. Teaching empathy to medical students: an updated, systematic review. Acad Med. 2013 Aug;88(8):1171-7. doi: 10.1097/ACM.0b013e318299f3e3. PMID 23807099
- [Background] Hojat M, Vergare MJ, Maxwell K, Brainard G, Herrine SK, Isenberg GA, Veloski J, Gonnella JS. The devil is in the third year: a longitudinal study of erosion of empathy in medical school. Acad Med. 2009 Sep;84(9):1182-91. doi: 10.1097/ACM.0b013e3181b17e55. PMID 19707055
- [Background] Griffith CH 3rd, Wilson JF. The loss of student idealism in the 3rd-year clinical clerkships. Eval Health Prof. 2001 Mar;24(1):61-71. doi: 10.1177/01632780122034795. PMID 11233586
- [Background] Haidet P, Dains JE, Paterniti DA, Chang T, Tseng E, Rogers JC. Medical students' attitudes toward patient-centered care and standardized patients' perceptions of humanism: a link between attitudes and outcomes. Acad Med. 2001 Oct;76(10 Suppl):S42-4. doi: 10.1097/00001888-200110001-00015. No abstract available. PMID 11597869
- [Background] Institute of Medicine (US) Committee on Quality of Health Care in America. Crossing the Quality Chasm: A New Health System for the 21st Century. Washington (DC): National Academies Press (US); 2001. Available from http://www.ncbi.nlm.nih.gov/books/NBK222274/ PMID 25057539
- [Background] Kim SS, Kaplowitz S, Johnston MV. The effects of physician empathy on patient satisfaction and compliance. Eval Health Prof. 2004 Sep;27(3):237-51. doi: 10.1177/0163278704267037. PMID 15312283
- [Background] Stacy R, Spencer J. Patients as teachers: a qualitative study of patients' views on their role in a community-based undergraduate project. Med Educ. 1999 Sep;33(9):688-94. doi: 10.1046/j.1365-2923.1999.00454.x. PMID 10476021
- [Result] Krupat E, Bell RA, Kravitz RL, Thom D, Azari R. When physicians and patients think alike: patient-centered beliefs and their impact on satisfaction and trust. J Fam Pract. 2001 Dec;50(12):1057-62. PMID 11742607
- [Result] Krupat E, Pelletier S, Alexander EK, Hirsh D, Ogur B, Schwartzstein R. Can changes in the principal clinical year prevent the erosion of students' patient-centered beliefs? Acad Med. 2009 May;84(5):582-6. doi: 10.1097/ACM.0b013e31819fa92d. PMID 19704190
- [Result] Krupat E, Rosenkranz SL, Yeager CM, Barnard K, Putnam SM, Inui TS. The practice orientations of physicians and patients: the effect of doctor-patient congruence on satisfaction. Patient Educ Couns. 2000 Jan;39(1):49-59. doi: 10.1016/s0738-3991(99)00090-7. PMID 11013547